CLINICAL TRIAL: NCT03240497
Title: The Influence of Breathing Techniques and Exposure to Cold on Inflammation During Human Endotoxemia, an Explorative Study'
Brief Title: Effects of Cold Exposure and Breathing Techniques on Immune Response
Acronym: EXPOCOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EXPOCOL
Record Dates: First submitted 2017-07-19; First posted 2017-08-07 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2017-07

CONDITIONS: Cold Exposure; Hyperventilation; Inflammation; Endotoxemia
MeSH Terms: conditions — Hyperventilation; Inflammation; Endotoxemia

STUDY DESIGN:
Intervention Model Description: A parallel randomized controlled explorative study in healthy male volunteers during experimental endotoxemia.
Who Masked: Outcomes Assessor
Masking Description: We employ a PROBE design (Prospective Randomized Open Blinded End-point) [41]. All subjects will receive a code number. Almost all of our end-points, especially the most important ones including the primary endpoint, are laboratory measurements, which will be performed blinded for the treatment of the subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cold Exposure (Experimental): A group of subjects (n=12) that will receive an extensive course in cold exposure similar in length to our previous study (total of 10 days) before the endotoxemia experiment.
  Interventions: Behavioral: Cold Exposure
- Strength Ventilation (Experimental): A group of subjects (n=12) that will be trained in the strength ventilation breathing technique before the endotoxemia experiment.
  Interventions: Behavioral: Strength Ventilation
- Cold Exposure and Strength Ventilation (Experimental): A group of subjects (n=12) that will receive both the cold exposure course (same as the STV group) as well as the training in the strength ventilation breathing technique (same as the CEX group) before the endotoxemia experiment.
  Interventions: Behavioral: Cold Exposure; Behavioral: Strength Ventilation
- Control group (No Intervention): A group of subjects (n=12) that will receive no training and will not be exposed to cold before the endotoxemia experiment.

INTERVENTIONS:
Behavioral: Cold Exposure — The start of the training is scheduled 7 to 12 days before the endotoxemia experiment day. Subjects in this group will participate in a 4 day intensive cold exposure course (see section 5.1). On day 1, venous blood will be sampled directly after ice water immersion. On day 4, venous blood will be sampled before the training procedures on that day and after the last ice water immersion.
  After the 4 day course, subjects will continue to practice cold exposure at home using cold showers. The timing and length of this training is analogous to the time spend on training in the cold in our previous study protocol [7].
  Arms: Cold Exposure; Cold Exposure and Strength Ventilation
Behavioral: Strength Ventilation — The training is scheduled 2 to 6 days before the endotoxemia experiment day. Subjects in this group will receive a detailed, written instruction about the strength ventilation technique (see section 5.1). In addition, they will receive a 2 hour instruction session during which the research team will supervise the practices and clarify the instructions of needed. Subjects are instructed not to practice the learned techniques at home.
  Arms: Cold Exposure and Strength Ventilation; Strength Ventilation

SUMMARY:
Inflammatory cytokines play a pivotal role in rheumatoid arthritis (RA) and innovative non-pharmacological therapies aimed at limiting cytokine production are highly warranted. Recently, our group showed that healthy volunteers trained in an intervention developed by 'Iceman' Wim Hof were able to voluntarily attenuate the pro-inflammatory response during experimental human endotoxemia (a model of systemic inflammation elicited by administration of lipopolysaccharide [LPS] in healthy volunteers). Subjects trained in the intervention exhibited profound increases in plasma adrenaline levels, a rapid increase of an anti-inflammatory cytokine and subsequent attenuation of the pro-inflammatory response.

The intervention consists of three elements, namely meditation, exposure to cold and breathing techniques. The meditation element is not likely to be involved. It was a very minor part of the training program and was not practiced during the endotoxemia experiments. Exposure to cold and the subsequent rewarming to normal body temperature may influence the inflammatory response through the release of immunomodulatory molecules like HSP-70. Also, exposure to cold can induce an ischemia-reperfusion-like state in the skin and peripheral tissue that is known to be involved in the downregulation of pro-inflammatory cytokines and upregulation of anti-inflammatory cytokines. The investigators anticipate that the third element, breathing techniques, is the major contributor to the anti-inflammatory effects of the intervention previously observed. The present study aims to explore the effects of the breathing technique ('strength ventilation'), the exposure to cold, and these two elements combined on the immune response during human endotoxemia. Elucidation of the relative contribution of the elements is of importance to establish a feasible, safe, and effective intervention for future use in patients.

Objective: The primary objective of the present study is to determine the effects of the 'strength ventilation' breathing technique and exposure to cold, both separately and in combination, on the inflammatory response during human endotoxemia. To this end, a 2 by 2 design will be employed. Additionally, an evaluation of the influence of the cold exposure and breathing technique on pain thresholds and oxygen tension in the mitochondria will take place.

DETAILED DESCRIPTION:
Auto-immune diseases are characterized by an inappropriate inflammatory response against tissues in the body. These diseases, of which rheumatoid arthritis (RA) is the most well-known, represent a major health care burden. Pro-inflammatory cytokines such as TNF-α, IL-6 and IL-1β are central in the pathogenesis of RA and many other auto-immune diseases. Biologics that antagonize inflammatory cytokines or their receptors, e.g. anti-TNF-α, soluble TNF-α-receptor, anti-IL-6 receptor, and IL-1 receptor antagonist, are very effective treatments. However, they are very expensive and can have serious side effects. Furthermore, the consequences of RA are currently completely beyond the patients' sphere of influence. Therefore, innovative therapies aimed at limiting inflammation in RA patients are warranted.

Recently, a study into the effects of an intervention developed by 'The Iceman' Wim Hof revealed that it is possible to voluntarily attenuate the pro-inflammatory response during experimental human endotoxemia (a standardized, controlled, and reproducible model of systemic inflammation elicited by administration of lipopolysaccharide (LPS) in healthy volunteers). The intervention developed by Hof consists of several elements, namely meditation, exposure to cold and breathing techniques. Subjects trained in this intervention exhibited profound increases in plasma adrenaline levels, a rapid increase of the anti-inflammatory cytokine IL-10, and subsequent attenuation of the pro-inflammatory response (e.g. plasma levels of TNF-α, IL-6, and IL-8) during experimental human endotoxemia. This intervention could therefore represent a treatment modality that would empower RA patients to exert self-control over their disease.

Based on these data, investigating the effectiveness of the intervention in RA patients is highly warranted. The study described in this protocol is part of a larger project in which the investigators ultimately strive to translate the intervention to clinical practice for RA patients. However, there are important issues that need to be addressed first. For example, feasibility and safety would be substantially improved if patients would only have to learn or practice one of the three elements of the intervention. The meditation element is not likely to be involved. It was a very minor part of the training program and was not practiced during the endotoxemia experiments. Also, there is no objective manner to measure this element and there is no hypothesis for a possible mechanism. Concerning the second element, exposure to cold, it would especially be of value to determine whether this element has additional value, because it is very demanding and might not be suitable for RA patients at all. The investigators anticipate that the third element, breathing techniques, is the major contributor to the anti-inflammatory effects of the intervention previously observed for reasons outlined below.

Breathing techniques First, although the healthy volunteers were trained in all three elements, subjects only practiced breathing techniques during the endotoxemia experiment. Second, the breathing techniques were characterized by cyclic hyperventilation, which has been shown before to result in increased adrenaline levels. Subjects practiced two types of breathing techniques during the endotoxemia experiment in our previous endotoxemia study. Both of these breathing techniques were characterized by cycles of hyperventilation. In one of the techniques (hyper/hypoventilation), subjects held their breath for up to several minutes after each hyperventilation period, while in the other technique (strength ventilation), subjects held their breath for only 10 seconds during which all muscles were tightened after each hyperventilation period.

Yet unpublished data (CMO 2014-1374) showed the effects of these two breathing techniques in the absence of cold exposure (or meditation) on plasma adrenaline levels. The investigators found these to be strongly correlated with the anti-inflammatory effects previously found. Both breathing techniques resulted in comparable increases in plasma adrenaline levels. Furthermore, adrenaline levels in subjects trained by Hof were comparable to those that were trained by an independent trainer previously not familiar with the intervention developed by Hof. Finally, adrenaline levels in subjects trained for 4 days were similar to those who were trained for only 2 hours.

Based on these results, it is hypothesized that the strength ventilation technique is the major contributor to the anti-inflammatory effects of the intervention previously observed. However, the effects of solely this breathing technique on the inflammatory response is not investigated yet. Furthermore, it cannot be ruled out that the exposure to cold has additional effects, since there are several ways in which exposure to cold could contribute to anti-inflammatory effects, as described below.

Exposure to cold First, exposure to cold and the subsequent rewarming to normal body temperature may influence the inflammatory response through the release of immunomodulatory danger associated molecular patterns (DAMP's), more specifically TLR-4 ligands such as heat shock protein 70 (HSP-70). It was shown that HSP-70 mRNA levels in isolated cardiac myocytes increased during rewarming after 2.5 hours of hypothermia. Furthermore, pre-incubation of human cells exposed to 4 °C for 1, 2, 3 and 4 hours induced synthesis and accumulation of HSP-70 upon recovery to 37 °C. The relevance of HSP-70 for the inflammatory response is evident from a study in which HSP-70 was shown to induce potent anti-inflammatory effects resembling induction of endotoxin tolerance in human monocytes.

Second, exposure to cold can induce an ischemia-reperfusion-like state in the skin and peripheral tissue. A study into the effects of cryotherapy showed that local cooling of the skin decreases local tissue perfusion. The combination of tissue hypoperfusion and reperfusion upon the reactive vasodilatation that follows after rewarming is a form of ischemia/reperfusion (I/R). The potency of I/R to protect tissue against ischemic damage is known as Ischemic Preconditioning (IPC). It has the potential to influence the immune response through several pathways. For instance, recent animal work has shown that I/R results in downregulation of pro-inflammatory cytokines such as TNF-α and IL-6 and upregulation of anti-inflammatory cytokines such as IL-10. Furthermore, hypoxia-inducible factor (HIF) has been shown to be a major contributor to the I/R-induced IL-10 response.

Third, exposure to cold could have a potentiating effect on the adrenaline release evoked by the breathing techniques. In a study of human volunteers, adrenaline levels were increased after 2 hours of sitting in a cold room. Interestingly, in a study during acute exercise in human volunteers, cold exposure prior to exercise was associated with an added immuno-stimulatory effect. Also, cytokineresponse of IL-1beta and IL-6 in ex vivo LPS-stimulated blood was lower in experienced ice-swimmers compared to inexperienced ice-swimmers.

Taken together, cold exposure may influence the in vivo response to endotoxemia. This might be mediated by direct, adrenaline-independent effects or by enhancing adrenaline levels elicited by strength ventilation.

Synthesis This study aims to explore the effects of two elements of the intervention initially developed by Hof, namely the strength ventilation breathing technique and the exposure to cold, on the immune response during human endotoxemia. Effects of both elements separately as well as in combination will be tested, the latter to explore the interplay between the elements.

In addition, an assesment will be made of the effects of the (combination of) breathing techniques and cold exposure on pain perception. In previous studies, trained subjects experienced substantially less flu-like symptoms during endotoxemia. This could be due to the attenuated immune response in these subjects, but also through other effects induced by the breathing techniques and/or cold exposure. To investigate this, quantitative sensory testing (QST) is used, an objective technique to measure pain thresholds.

Finally, non invasive measurements of oxygen tension in the mitochondria will be used to asses mitochondrial function during human endotoxemia by using the Protoporphyrin IX-Triplet State Liftime Technique (PpIX-TSLT).

Mitochondrial dysfunction is an important element in the pathophysiology of sepsis. However, a valid non-invasive method to measure mitochondrial function is not yet available. In animal models, the PpIX-TSLT technique has shown to be a feasible technique to measure alterations in mitochondrial oxygen tension during endotoxemia. This has never been studied in humans during endotoxemia. Furthermore, the exposure to cold and especially the breathing technique may influence oxygen tension in the mitochondria as well, as blood gas parameters (e.g. pCO2, acid base balance etc.) fluctuate to a large extent during the practicing of this technique.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male
* Healthy

Exclusion Criteria:

* Prior experience with any of the elements of the intervention developed by Hof
* Prior experience with other breathing, meditation, or cold exposure techniques
* Prior experience with mindfulness or yoga
* Prior experience with exposure to cold showers
* Frequent visits to sauna facilities (more than 1/month)
* Use of any medication
* Smoking
* History of asthma
* History of porphyria
* Previous spontaneous vagal collapse
* History of atrial or ventricular arrhythmia
* (Family) history of myocardial infarction or stroke under the age of 65 years
* Cardiac conduction abnormalities on the ECG consisting of a 2nd degree atrioventricular block or a complex bundle branch block
* Hypertension (defined as RR systolic > 160 or RR diastolic > 90)
* Hypotension (defined as RR systolic < 100 or RR diastolic < 50)
* Renal impairment (defined as plasma creatinin >120 μmol/l)
* Liver enzyme abnormalities
* Medical history of any disease associated with immune deficiency
* CRP > 20 mg/L, WBC > 12x109/L, or clinically significant acute illness, including infections, within
* 4 weeks before endotoxin administration
* Participation in a drug trial or donation of blood 3 months prior to the LPS challenge
* Use of recreational drugs within 7 days prior to endotoxemia experiment day
* Recent hospital admission or surgery with general anaesthesia (<3 months)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
circulating TNF-α | 8 hours
  The main study endpoint is the difference in circulating TNF-α over time following LPS administration between groups

SECONDARY OUTCOMES:
Cytokines | 8 hours
  Levels of other circulating cytokines (including, but not limited to IL-6, IL-10 and IL-1RA)
Plasma adrenaline levels | 8 hours
  routine analysis methods also used for patient samples (high-performance liquid chromatography with fluorometric detection
Plasma cortisol levels | 8 hours
  routine analysis methods also used for patient samples performed by the Department of Laboratory Medicine of the Radboud University Nijmegen Medical Centre.
- Blood gas parameters | 8 hours
  Blood gas parameters will be analyzed using the i-STAT Blood Gas Analyzer (Abbot, Hoofddorp, The Netherlands).
- Mitochondrial oxygen tension | 8 hours
  The COMET device measures cutaneous mitochondrial oxygen tension (MitoPO2) over time. MitoPO2 is measured by means of delayed fluorescence of mitochondrial protoporphyrin IX (PpIX) [6]. Microcirculatory flow can be stopped by applying pressure with the measuring probe on the skin, enabling the determination of the oxygen disappearance rate (ODR)
- Metabolome | 8 hours
  The metabolome will determined using the 'Kenkodo @home' sampling set, developed by Metabolomic Discoveries GmbH (http://www.metabolomicdiscoveries.com/).
  Using a minimally invasive finger prick we will obtain 10µl (microliter) of blood from the subjects. The used Mitra Sampling Device is a Class 1 medical device (D254956) and complies with FDA good manufacturing practices. Samples will be analyzed at Metabolomic Discoveries GmbH.
- Body temperature | 8 hours
  The course of body temperature will be determined every 30 minutes for the first 8 hours after endotoxine administration using an infrared tympanic thermometer (Sherwood Medical, 's-Hertogenbosch, the Netherlands).
- Illness score | 8 hours
  To monitor the onset and alterations of endotoxine-induced symptoms, all subjects will be asked to score the severity of nausea, headache, shivering, muscle- and backpain every 30 minutes during the course of the experiment. Symptoms are scored on a scale ranging from 0 (symptom not present) to 5 (symptom is worst ever experienced).
heart rate | 8 hours
  Heart rate will be continuously measured by connecting the arterial catheter to an arterial pressure monitoring set. Data will be recorded from the patient monitor every 30 seconds by a custom in-house-developed data recording system.
Blood pressure | 8 hours
  Blood pressure will be continuously measured by connecting the arterial catheter to an arterial pressure monitoring set. Data will be recorded from the patient monitor every 30 seconds by a custom in-house-developed data recording system.
- Leukocyte counts and differentiation | 8 hours
  Measurements of haemoglobin, leukocyte and thrombocyte count, determinations of kidney and liver function, amylase, CRP, cortisol and catecholamines will be performed by the laboratory for clinical chemistry at the Radboud university medical center.
Pain thresholds: PPT | 8 hours
  PPT will be measured on the left and right bodyside once at three locations. Single pulse evoked pain measurement is performed by one pulse at 150% of the EPT and assessed on a VAS. .
Pain thresholds: EPTT | 8 hours
  Electrical Pain Tolerance Thresholds (EPTT) (test stimulation) are assessed and expressed in milli-Ampère on the m. Rectus femoris contralateral to the dominant hand
- Presence of TLR ligands in plasma | 8 hours
  HSP70 will be measured in using ELISA. Presence of other TLR ligands in plasma will be studied using transfected HEK-blue TLR cells (Invivogen).
- HSP70 levels in plasma. | 8 hours
  HSP70 will be measured in using ELISA. Presence of other TLR ligands in plasma will be studied using transfected HEK-blue TLR cells (Invivogen).
- Production of inflammatory mediators by ex vivo-stimulated leukocytes | 8 hours
  Ex vivo leukocyte stimulation by different pathogens will be performed at the Laboratory of General Internal Medicine of the Radboud university medical center. Cytokines in supernatants of stimulated leukocyte cultures will be determined by ELISA. Inflammatory transcriptional pathways will be determined by quantitative PCR/microarrays/RNA sequencing at the Laboratory of General Internal Medicine of the Radboud university medical center and/or the University of Groningen medical center.
- Inflammatory transcriptional pathways sequencing | 8 hours
  by use of qPCR/microarrays/RNA

CONTACTS AND LOCATIONS:
Overall Officials: Jelle Zwaag, MSc, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Centre, Intensive Care, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wefers Bettink MA, Zwaag J, Schockaert B, Pickkers P, Kox M, Mik EG. Measuring mitochondrial oxygenation and respiration during systemic inflammation in humans in vivo. Sci Rep. 2025 Jul 16;15(1):25815. doi: 10.1038/s41598-025-10715-6. PMID 40670486
- [Derived] Zwaag J, Naaktgeboren R, van Herwaarden AE, Pickkers P, Kox M. The Effects of Cold Exposure Training and a Breathing Exercise on the Inflammatory Response in Humans: A Pilot Study. Psychosom Med. 2022 May 1;84(4):457-467. doi: 10.1097/PSY.0000000000001065. Epub 2022 Feb 23. PMID 35213875